CLINICAL TRIAL: NCT01371279
Title: EvaluAtion of Predictive Value of Multisite Intracardiac EchoCardiography During Imaging of Structure and funCTION of Left Atrial Appendage in Comparison to Transesophageal Echocardiography
Acronym: ActionICE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre of Postgraduate Medical Education (Other)
Responsible Party: Sebastian M.Stec / Jakub Baran, Medical Centre of Postgraduate Education, Poland
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1-Stec
Record Dates: First submitted 2011-05-23; First posted 2011-06-10 (Estimated); Last update posted 2011-06-17 (Estimated); Status verified 2011-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Intra-Cardiac Echocardiography guided atrial fibrillation ablation — 8-F or 10-F phase array ICE-probe
  Other Names: AcuNav Siemens Ag Medical Solution

SUMMARY:
This is a 2- component, single center study, witch aims to evaluate the efficacy of multisite intracardiac echocardiography (mICE) imaging of left atrial appendage (LAA) and in detecting thrombus located in LAA as compared to transesophageal echocardiography (TEE). The study group will consist of patients eligible for atrial fibrillation (AF) ablation procedure (Component I) or cardioversion (Component II).

First component will enroll 100 patients; these patients will undergo clinically indicated TEE & cardiac catheterization procedures with ICE(AF ablation). Second component will enroll 15-20 patients with AF or atrial flutter in whom a thrombus in LAA was detected by TEE prior to electrical cardioversion. The ICE probe will be located in multiple positions in the right atrium (RA), coronary sinus (CS), pulmonary artery (PA), right ventricular outflow tract (RVOT) and esophagus. This will enable the investigators to compare sensitivity and specificity of mICE and TEE.

This study will examine two hypotheses in AF patients undergoing invasive cardiac procedures:

Hypothesis 1: That ICE has comparable efficacy to TEE in visualization of LAA from multiple positions (RA,CS,PA,RVOT and esophagus ). This will be evaluated during the component I of the study.

Hypothesis 2: That ICE can identify low risk patients, CHADS Score < 2,0 in whom immediate cardioversion during the procedure is as safe as based on conventional strategy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with paroxysmal/persistent AF
2. Patients with or without structural Heart Disease.
3. Men or Women aged 18 years or older.
4. Patients undergoing an invasive catheterization procedure including right heart catheterization.
5. Patients who give an informed consent for participation in the study.
6. Patients who have undergone a trans-esophageal echocardiogram within the last 48 hours. Patient witch CHADS2 score > 2

Exclusion Criteria:

1. Patients in whom placement of an ICE catheter for adequate atrial visualization is technically not feasible (Right atrium or Esophagus).
2. Women of child bearing potential, in whom pregnancy cannot be excluded.
3. Patients with any medical condition or social circumstance, which in the opinion of the investigator, would make the patient's successful completion of the study doubtful

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-06; Primary Completion 2013-02 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Predictive value of ICE compared to TEE in visualisation of morphology and thrombus in LAA. | intraoperative - up to six hours
  Predictive value of ICE compared to TEE in visualization of morphology (area and volume of LAA) and function of LAA (emptying velocity and ejection fraction of LAA) - offline analyses will be conducted. Quality of LAA imaging will be assessed using 5-grade scale, and compared to that obtained by TEE. Grade 0 means unacceptable quality wheras grade 5 means exellent view of LAA. Exclusion of existence of thrombus in LAA by mICE will enable electrical cardioversion of AF during AF ablation procedure. That will by assessed using binary scale - YES or NO.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Postgraduate Medical School, Grochowski Hospital, Grenadierow 51/59, Warsaw, Poland

REFERENCES:
- [Derived] Baran J, Stec S, Pilichowska-Paszkiet E, Zaborska B, Sikora-Frac M, Krynski T, Michalowska I, Lopatka R, Kulakowski P. Intracardiac echocardiography for detection of thrombus in the left atrial appendage: comparison with transesophageal echocardiography in patients undergoing ablation for atrial fibrillation: the Action-Ice I Study. Circ Arrhythm Electrophysiol. 2013 Dec;6(6):1074-81. doi: 10.1161/CIRCEP.113.000504. Epub 2013 Nov 15. PMID 24243787